CLINICAL TRIAL: NCT01237392
Title: Ultrasonic Surgical Wound Debridement vs. Standard Sharp Debridement In the Treatment of Chronic Wounds: A Single Center, Randomized, Parallel, Clinical Outcome Trial
Brief Title: Ultrasonic Wound Debridement vs. Standard Sharp Debridement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calvary Hospital, Bronx, NY (Other)
Responsible Party: Principal Investigator, Oscar M. Alvarez, PhD, Director, Center for Curative and Palliative Wound Care, Calvary Hospital, Bronx, NY
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NYSDH-Dbr-06-08
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Skin Ulcers
Keywords: wound debridement; requiring debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contact Ultrasonic Debridement Device (Active Comparator)
  Interventions: Device: Contact ultrasonic debridement device
- Standard Sharp Debridement (Active Comparator)
  Interventions: Device: Contact ultrasonic debridement device

INTERVENTIONS:
Device: Contact ultrasonic debridement device — Cavitational ultrasound wound debridement device
  Other Names: SonicOne, Misonix Inc, Farmingdale NY

SUMMARY:
A single center, randomized, parallel, clinical outcome trial to compare the rate of healing in chronic wounds debrided with either high energy ultrasonic debridement (with cavitation) or standard of care sharp debridement.

ELIGIBILITY:
Inclusion Criteria:

* Chronic wound needing debridement >3 cm2
* Ulcer history >4mo
* Adequate arterial blood flow (ABI>0.7)
* Venous, Inflammatory, Pressure, Diabetic

Exclusion Criteria:

* Bleeding disorder
* ABI<0.7
* Uncontrolled diabetes
* Taking systemic corticosteroids
* Chemotherapy
* Participating in another study
* Treatment with Apligraft, Dermagraft, or Regranex within 90 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Time to complete wound closure | 12 and 24 weeks

SECONDARY OUTCOMES:
Relative rate of wound healing | 8, 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar M Alvarez, PhD, Principal Investigator — Director, Wound care Center, Calvary Hospital; Martin E Wendelken, DPM, RN, Study Director — Physician, Wound Care Center, Calvary Hospital
Locations (1):
- Calvary Hospital Center for Curative and Palliative Wound Care, The Bronx, New York, United States